CLINICAL TRIAL: NCT00451438
Title: Investigation of Muscle Activity Pattern of Gluteus Medius and Tensor Fascia Lata in Patients With PFPS
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 200701003R
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2007-01

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; electromyography; gluteus medius; tensor fascia lata
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the muscle activity of gluteus medius and tensor fascia lata in health control group and patients with PFPS during submaximal isometric muscle contraction.The research question :Is there any difference of muscle activity of gluteus medius and tensor fascia lata between health control group and patients with PFPS during submaximal isometric muscle contraction ？Null hypothesis:There is no difference of muscle activity of gluteus medius and tensor fascia lata between health control group and patients with PFPS during submaximal isometric muscle contraction.

DETAILED DESCRIPTION:
Basic data

- Name, age, sex, BW, BH, pain VAS scale（VAS-activity）, affected side, dominate leg, symptom duration, activity level

Measurement

* Flexibility of iliotibial band：Ober test
* EMG data collection during 8s submaximal muscle contraction
* Muscle strength measurement of hip abductors

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years old
* Insidious onset of symptoms
* Pain exist at least 3 month, VAS activity>4
* Two of the following activities induce pain at anterior or retropatellar site prolonged sitting, stair-climbing, squatting, running, kneeling, and hopping/jumping
* Diagnosed by an orthopedic surgeon

Exclusion Criteria:

* History of lower extremity fracture or operation
* Neurological disease involved
* Observed knee deformity
* Other well-defined musculoskeletal problems in lower extremity

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2007-01; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwa Jan, Master, Study Chair — NTU department of physical therapy